CLINICAL TRIAL: NCT02416843
Title: Metabolic and Immune System Responses to a Mixed Meal in Human Adipose Tissue and the Circulation
Brief Title: Metabolic and Immune System Responses to a Mixed Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Unilever R&D (Industry)
Responsible Party: Principal Investigator, Rebecca Travers, PhD Student, University of Bath
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11/SW/0193
Record Dates: First submitted 2015-04-01; First posted 2015-04-15 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Inflammation
Keywords: Adipose tissue; metabolism; inflammation; post-prandial; human
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lean (Experimental): Consumption of a mixed meal relative to individual resting metabolic rate.
  Interventions: Other: Consumption of a mixed meal
- Overweight (Experimental): Consumption of a mixed meal relative to individual resting metabolic rate.
  Interventions: Other: Consumption of a mixed meal
- Obese (Experimental): Consumption of a mixed meal relative to individual resting metabolic rate.
  Interventions: Other: Consumption of a mixed meal

INTERVENTIONS:
Other: Consumption of a mixed meal — Participants will consume a mixed meal and postprandial responses in blood and adipose tissue will be investigated over 6 hours and compared to baseline.

SUMMARY:
Overweight and obesity are major problems and their complications such as cardiovascular disease and type 2 diabetes mellitus pose great burdens on healthcare systems. There is accumulating evidence to support obesity being a chronic inflammatory disorder mediated in part by the expansion of adipose (fat) tissue.

Knowledge of the role of adipose tissue itself has changed dramatically and it has emerged that in addition to storing energy as fats; adipose tissue secretes and responds to various chemical messengers in the body that are related to metabolism and inflammation. After a meal has been consumed, changes in metabolic (and some inflammatory) markers are seen in the blood, which may be influenced by metabolic and inflammatory changes occuring in the adipose tissue itself.

The investigators therefore plan to investigate these changes in adipose tissue before and after a meal and compare them to changes occurring in the blood. They also plan to investigate whether these responses are different in people who are overweight compared to 'normal' weight.

Participants will include males aged between 35-55 years who fit the criteria for inclusion. After taking some preliminary measurements and monitoring of normal daily activities, participants will attend one day of Laboratory testing in the Physiology Laboratories at the University of Bath.

By investigating differences in metabolism and inflammation in adipose tissue and the circulation it is hoped that more will be learnt about the development of diseases associated with being overweight and ultimately help to develop more effective methods for prevention and treatment.

DETAILED DESCRIPTION:
The aim of this research is to investigate differences in metabolism and inflammation in adipose tissue and the circulation in response to a meal with increasing adiposity. It is hypothesised that participants with increased fat mass, will have a more pronounced inflammatory response to a meal compared to participants with a 'healthy' weight. The inflammatory response will be assessed by measuring changes in gene expression and protein secretion in the adipose tissue and by measuring markers of metabolism, insulin resistance, cardiovascular disease and inflammation in the blood.

Following advertisement of the study, interested potential participants will be asked to contact the Chief Investigator for further information via email/telephone correspondence. There will be an initial assessment of eligibility based on inclusion/exclusion criteria and, if these requirements are met, the potential participant will be invited to a meeting to further discuss the trial. After they have read the participant information sheet and seen the flowchart outlining the timeline for the study, if they would like to take part, they will be asked to sign a consent form. Dates will then be scheduled for some preliminary anthropometric measurements to be taken, 9 days of physical activity monitoring and the trial date (1 full day in the laboratory only).

Preliminary measurements:

Preliminary testing will include anthropometric measurements of height, weight, waist and hip circumferences, sagittal waist height and blood pressure. These measurements will take place at the University of Bath Physiology Laboratories.

Physical activity monitoring:

For 9 days, participants will be fitted with a physical activity monitor (Actiheart™) and asked to record a corresponding diary of their physical activity during this period to aid its interpretation and allow a more accurate calculation of average daily activity energy expenditure. Participants should not make any conscious changes to their normal lifestyle habits/routines during this period. The first 2 days of activity monitoring will be excluded from analysis to account for reactivity.

Main trial day:

In the 3 days prior to the main trial day, participants will be asked to record their food and drink intake and 48 hours before they should refrain from performing any strenuous physical activity. In the 24 hours prior participants should also refrain from consuming any alcohol or caffeine.

Participants should arrive at the Sports Training Village, University of Bath in the morning following a 10 hour fast where they will have their body composition precisely assessed using a dual-energy Xray absorptiometer (DEXA). They will then be taken to the Physiology Resting Laboratory where baseline expired gases will be collected for assessment of resting metabolic rate (RMR). A cannula will be inserted into a forearm vein and baseline blood sample(s) taken for analysis of metabolic/inflammatory markers and isolation of T cells. A fat sample will also be obtained using a needle aspiration technique.

The participant will then be asked to consume a breakfast type meal that is high in carbohydrate and fat contents consisting of brioche, jam, butter, and milkshake which has been adapted from a meal used by Rijkelijkhuizen J. et al, 2008, which induced stronger beta cell responses (i.e. of insulin) compared to a glucose load and showed differences with insulin sensitivity, so this meal type should identify differences in metabolism based on adiposity.

Furthermore, there is some evidence that high starch/low fibre foods may induce greater inflammation (Manning, Sutherland et al. 2008). The meal composition for all individuals will be identical but the energy content from carbohydrate will be calculated as a portion of the individuals' resting metabolic rate. This allows standardisation of energy intake for differences body weight/composition and will reflect energy requirements of the individual whilst at rest.

The meal should be consumed within 15 minutes and blood samples will be taken from the cannula at 15, 30, 60, and 90 minutes and then at every hour for 6 hours after consumption of the meal to monitor changes in metabolic and inflammatory markers. Additional blood samples will be obtained at 2 and 6 hours post meal by venepuncture for analysis of inflammatory markers as there is evidence that the cannula can stimulate local inflammation which interferes with the true result.

Expired gas samples for RMR will also be taken hourly and indirect calorimetry will be used to estimate relative fat and carbohydrate metabolism in response to the meal.

A second fat sample will be taken at 6 hours to examine inflammatory and metabolic responses to the meal within adipose tissue. A second blood sample for T cell isolation will also be obtained at this time point to examine corresponding metabolic/inflammatory responses in T cells.

Analysis:

On the day of the trial whole blood will be analysed for white blood cell count, glucose and lactate. Plasma and serum samples will be extracted from the whole blood via centrifugation and stored at -80. Monocytes and T lymphocytes (populations of white blood cells) will also be isolated from whole blood for later assessment of insulin sensitivity and culture experiments.

In each fat sample, separate portions of either adipose tissue or adipocytes (isolated from the other cells within the adipose tissue using a digestion method) will be cultured and media collected for later investigations. mRNA expression will also be examined in adipose tissue and isolated adipocytes. The remaining cells from the adipose tissue (SVF) will also be stored for later analysis of cell populations using flow cytometry, and expression/secretion analysis.

ELIGIBILITY:
Inclusion Criteria:

Subjects should be:

* Nonsmokers
* Weight stable for more than 3 months

Exclusion Criteria:

Subjects should not :

* have a personal history of/existing cardiovascular disease, metabolic disease or dyslipidaemia
* be taking medications that may influence lipid or carbohydrate metabolism
* have food intolerances/allergies to any component of the meal (i.e. dairy or wheat)
* Perform no more than 6 hours of strenuous physical activity or 10 hours of moderate intensity physical activity per week (as these individuals will not fit the meal standardisation procedure)

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes in IL6 mRNA expression in adipose tissue | 6 hours
  mRNA expression of IL6 will be measured in adipose tissue samples obtained pre and 6 hours post consumption of the mixed meal to assess for postprandial inflammatory changes in adipose tissue.

SECONDARY OUTCOMES:
Changes in IL-6 secretion by adipose tissue | 6 hours
  Adipose tissue explants will be cultured for 3 hours using samples obtained before and 6 hours after the meal to assess for any changes in IL-6 secretion.
Analysis of insulin stimulated pathways | 6 hours
  Activation/inhibition of insulin stimulated pathways in isolated adipocytes (by assessment of Akt/IRS1 phosphorylation by western blot analysis) will be assessed before and 6 hours after the meal.
Characterisation of immune cell populations in adipose tissue | 6 hours
  Adipose tissue samples will be examined for their resident immune cell populations and compared to those in blood and characterised according to their respective activation statuses, in particular CD4+ and CD8+ T lymphocytes using flow cytometry analysis.
Effect of adipocytes on T Lymphocyte activation | 6 hours
  To examine whether adipocytes influence T lymphocyte function/ability to activate (following stimulation) before and after a meal by culture/stimulation of isolated T cells with their own adipocyte culture media pre and post - meal (analysis of proliferation and activation by flow cytometry).

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Thompson, PhD, Principal Investigator — University of Bath; James A Betts, PhD, Principal Investigator — Univeristy of Bath; Alexandre C Motta, PhD, Principal Investigator — Unilever R&D; Rebecca L Travers, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath - Department for Health, Bath, Bath and North East Somerset, United Kingdom